CLINICAL TRIAL: NCT03369119
Title: Phase 4 Study of Oral Montelukast Hospitalized Preschool Children
Brief Title: Effect of Addition Oral Montelukast to Standard Treatment in Acute Asthma in Hospitalized Preschool Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, Pediatric Allergy Specialist, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.10.0.İEG.0.11.00.01/003247
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Acute Asthma; Acute Wheezy Bronchitis
Keywords: Acute asthma; Montelukast; Hospitalized children; Preschool children
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast (Active Comparator): Children received 4 mg oral montelukast granule daily until discharge.
  Interventions: Drug: Montelukast 4 Mg Oral Granule
- Placebo (Placebo Comparator): Children receive 4 mg oral placebo montelukast granule daily until discharge
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Montelukast 4 Mg Oral Granule
  Other Names: Montelukast sodium
  Arms: Montelukast
Drug: Placebos
  Arms: Placebo

SUMMARY:
Leukotriene receptor antagonists (LTRAs) are well established in the management of outpatient asthma. Montelukast is a potent, specific, orally active, cysteinyl leukotriene receptor antagonist with a rapid onset of action.However, there is very little information as to their role in acute asthma exacerbations.

The purpose of this study is to determine if adding oral montelukast to the maximal standard treatment in children hospitalized for acute asthma has any additive benefit.

DETAILED DESCRIPTION:
Background: Montelukast is a potent, specific, orally active, cysteinyl leukotriene receptor antagonist with a rapid onset of action.

Objective: To evaluate the effect of the addition of a single dose of oral montelukast to standard therapy in acute asthma. Design: Double-blind, randomised, controlled, parallel group trial. Setting: Pediatric service of Education and training Hospital Patients: Children with the ages of 6-60 months who were hospitalized for acute asthma Intervention: Children received montelukast 4 mg or placebo orally in addition to the standard therapy. Clinical asthma score was recorded before administering study medication and thereafter, 4 hourly until discharge. Main outcome measure: The primary outcome was discharge rates.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of at least 4 wheezing attacks
* Children with the ages of 6-60 months
* Children whose parents accept to give written informed consent

Exclusion Criteria:

* Chronic diseases (e.g. malnutrition, anatomic malformation of the respiratory tract, chronic lung or heart disease, gastroesophageal reflux disease and cystic fibrosis)
* Children with a history of chronic drug use (e.g. antiepileptics and immune suppressives)

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | within the 5 days from hospitalization
  The primary outcome was the difference in mean length of hospital stay as an hour between the 2 groups.

SECONDARY OUTCOMES:
Difference in clinical asthma score | Within 72 hours from hospitalization
  Improvement of clinical asthma scores between the 2 groups within 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cem H. Razi, M.D., Principal Investigator — Pediatric Allergy Specialist
Locations (1):
- Kecioren Education and Training Hospital, Ankara, Keçiören, Turkey (Türkiye)